CLINICAL TRIAL: NCT06126744
Title: The PuMP Trial: "A Multistage Phase 1 Open-Label Study to Evaluate the Safety, Tolerability and Efficacy of the Oncolytic HSV1 MVR-C5252 in Patients With Recurrent High-Grade Glioma"
Brief Title: Open-Label Study to Evaluate the Safety, Tolerability and Efficacy of the Oncolytic HSV1 MVR-C5252
Acronym: PuMP
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Principal Investigator, Mustafa Khasraw, MBChB, MD, FRCP, FRACP, Professor of Neurosurgery, Duke University
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: Pro00112883
Record Dates: First submitted 2023-09-24; First posted 2023-11-13 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Recurrent High Grade Glioma
MeSH Terms: conditions — Glioma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- MVR-C5252 (Experimental): Open label single arm infusion of MVR-C5252, genetically engineered type 1 oHSV (oncolytic herpes simplex viruses) into the tumor via Convection-enhanced delivery (CED) a modality that can bypass the BBB (Blood Brain Barrier), allowing the intracranial delivery through the BBB and avoiding systemic toxicities.
  Interventions: Biological: MVR-C5252

INTERVENTIONS:
Biological: MVR-C5252 — MVR-C5252 is a genetically modified next generation oncolytic herpes simplex virus 1 (oHSV1) with an active domain of human IL-12 and Fab fragment of anti-PD-1 antibody. This is a Phase 1 open label study designed to determine the safety and tolerability of MVR-C5252. The dose-escalation portion of the study will be conducted in 4 stages to evaluate the safety of infusion and determination of the MTD/RP2D followed by efficacy assessment.

SUMMARY:
This is a Phase 1 open label study designed to assess the safety and tolerability of the oncolytic herpes simplex virus 1 (oHSV1) study drug, MVR-C5252, administered intratumorally by convection-enhanced delivery (CED) in patients with recurrent high-grade glioma. Once the safety and maximum tolerated dose (MTD) is established in the dose escalation portion of the trial, a dose expansion cohort at the recommended phase 2 dose (RP2D) in patients with isocitrate dehydrogenase (IDH) wildtype recurrent glioblastoma (GBM) will evaluate preliminary efficacy of the study drug.

DETAILED DESCRIPTION:
Oncolytic HSV1 (oHSV1) was the first viral vector studied in clinical trials to treat malignant glioma with positive outcomes for tolerability and potential clinical benefits. MVR-C5252 is a genetically modified next generation oHSV1 with an active domain of human IL-12 and Fab fragment of anti-PD-1 antibody. During viral replication, IL-12 and anti-PD-1 antibody are expressed and secreted into the tumor microenvironment, acting synergistically by increasing the T cell infiltration, converting the cold (immune suppressing) tumor to hot (immune active) tumor, and inducing anti-tumor specific immunity. This study is investigating if oHSV1 MVR-C5252 administered via CED can overcome the BBB (Blood Brain Barrier) in patients with recurrent high-grade glioma. This study will enroll patients in 4 Stages. In Stage 1, externalized Synchromed II pump will be used to deliver Gadoliunium followed by MVR-C5252 for a single administration on Day 1. Stage 2, two infusions will be administered-on days 1 and 28 via the internalized pump. For patients accrued on Stage 3, the second infusion of study drug (Cycle 1, infusion 2) will occur 7 ± 1 days after 1st infusion for a total of 6 cycles (12 infusions). Stage 4, the dose expansion portion of the study, will commence once a MTD/RP2D is established. Within Stage 4 the efficacy of the study drug, as measured by progression-free 6 months survival will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. Age >18 years of age
2. Disease recurrence of at least 1x1cm and a maximum of 3x3cm of enhancing tumor:

   Dose escalation portion: patients with recurrent high-grade glioma, IDH wt or IDH mutated, grade 3 or grade 4 based on imaging.

   Dose expansion portion: Recurrent, IDH wt, glioblastoma, WHO grade 4. Diagnosis has be made using the 2021 WHO Classification of Tumors of the CNS.
3. The neurosurgeon must confirm (a) the tumor location (> 1 cm from eloquent brain), (b) that the placement of infusion catheter within or through the progressive enhancing tumor is feasible and is at a safe distance to eloquent brain function. These aspects will be determined prior catheter placement on the basis of prior (screening) MRI and then at the time of catheter placement on the basis of a CT scan prior to infusion. The tip of the catheter must be placed as follows:

   1. Within the enhancing portion or in the vicinity of enhancement of target lesion (i.e., infiltrative disease)
   2. ≥ 0.5 cm from ventricles
   3. ≥ 1 cm deep into the brain
   4. ≥ 0.5 cm from the corpus callosum
4. If a histological or pathological confirmation of recurrence (< 6 weeks) is not available, a pre-infusion biopsy will be required to confirm recurrence.
5. Adequate pulmonary function, with a baseline pulse oximetry of at 90% on room air.
6. The subject must have received standard radiation therapy plus temozolomide and be refractory to radiation therapy plus temozolomide prior to enrollment.
7. Prior to administration of MVR-C5252, the presence of recurrent tumor must be confirmed by histopathological analysis. (Distinguishing between recurrent active tumor and radiation necrosis is important to avoid delivering MVR-C5252 when there is no active disease).

   Should participants have further surgical resection at any time following their participation in the study, patients will be invited to make any biospecimens available for correlative research.
8. Karnofsky Performance Status (KPS) ≥ 70%
9. Labs:

   1. platelets ≥ 100,000 unsupported at initial screening, but ≥ 125,000 supported prior to biopsy/catheter insertion
   2. hemoglobin ≥ 9 gm/dL, ANC ≥ 1000/µL
   3. creatinine ≤ 1.5x upper limit of normal (ULN)
   4. total bilirubin ≤ 1.5 x ULN, AST/ALT ≤ 2.5 x ULN (subjects with known or suspected Gilbert's syndrome are excluded if total bilirubin > 3.0 x ULN or direct bilirubin > 1.5 x ULN)
   5. PT, aPTT ≤ 1.2 x ULN prior to biopsy (if patient is taking warfarin, INR should be obtained and be < 2.0)
10. Able to undergo MRI brain with and without contrast
11. If the patient is a sexually active female of childbearing potential, whose partner is male, or if the patient is a sexually active male, whose partner is a female of child bearing potential, the patient must use appropriate contraceptive measures for the duration of the treatment and for 6 months afterwards. Female patients of childbearing potential must have a negative serum pregnancy test at the time of screening and within 48 hours of starting the MVR-C5252 infusion.
12. Signed informed consent approved by the Institutional Review Board

Exclusion Criteria:

1. Prior, unrelated malignancy requiring current active treatment with the exception of cervical carcinoma in situ and adequately treated basal cell or squamous cell carcinoma of the skin
2. Patients who are pregnant or breastfeeding
3. Patients with contrast-enhancing tumor crossing the midline, multifocal tumor, infratentorial tumor, tumor in eloquent brain regions, extensive tumor dissemination (subependymal or leptomeningeal), or in unsafe brain regions per the opinion of the treating neurosurgeon
4. Unstable systemic disease in the opinion of the treating physician.
5. Active infection requiring systemic therapy or causing fever (temperature > 38.1˚C) or subjects with unexplained fever (temperature > 38.1˚C) within 7 days prior to the day of investigational product administration.
6. Patients on >4 mg per day of dexamethasone within the 2 weeks prior to admission for MVR-C5252 infusion or systemic therapy with immunosuppressive agents within 28 days prior to admission for MVR-C5252 infusion
7. Patients who have not completed standard of care treatment prior to participation in this trial
8. Less than 12 weeks from radiation therapy, unless progressive disease outside of the radiation field or 2 progressive scans at least 4 weeks apart or histopathologic confirmation of recurrent tumor
9. Treated with immunotherapeutic agents prior to MVR-C5252 treatment, within 4 weeks, alkylating agents within 4 weeks, nitrosoureas within 6 weeks, or non-alkylating chemotherapy within 2 weeks before enrollment, unless the patient has recovered from the expected toxic effects of such therapy
10. Treated with antiangiogenic agents (i.e., bevacizumab) within 4 weeks before biopsy
11. Patients who require an attenuated or live vaccine within 28 days prior to the first trial drug administration and during the study treatment period
12. Prior treatment with any oncolytic virus, cell therapy or gene therapy.
13. Prior antitumor treatment with intracranial implants, such as Carmustine
14. Previous history of allergic reactions to similar biological components such as HSV-1, IL-12 or anti-PD-1 antibodies, or with known allergic reactions to any component of the MVR-C5252 prescription, including glycerol.
15. Systemic use (other than topical) of anti-HSV drugs (including, but not limited to, acyclovir, valaciclovir, penciclovir, famciclovir, ganciclovir, foscarnet, cidofovir, etc.)
16. Patients with cardiac risks including congestive heart failure (as defined by New York Heart Association Functional Classification III or IV), unstable angina, serious uncontrolled cardiac arrhythmia, a myocardial infarction within 6 months prior to study entry, or a history of myocarditis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Estimated)
Dates: Start 2024-06-11 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Stage 1: Proportion of patients with dose-limiting toxicity (DLT) during the single infusion | Day 1 of treatment until 28 days post first infusion
  Proportion of patients with dose-limiting toxicity (DLT) during the single infusion
Stage 2: Proportion of patients with dose-limiting toxicity (DLT) during 2 infusions using the internalized Ascenda catheter | Day 1 of treatment until 28 days post second infusion for a total of up to 56 days post first infusion
  Proportion of patients with DLT who have received two infusions on days 1 and 28
Stage 3a: Proportion of patients with dose-limiting toxicity (DLT) after each cycle with two infusions on days 1 and 8 | Day 1 of treatment until 28 days post second infusion for a total of up to 35 days post first infusion
  Proportion of patients with DLT who have received two infusions on days 1 and 8
Stage 3b: Determine the MTD/RP2D | Day 1 of treatment until 28 days post second infusion for a total of up to 35 days post first infusion for all the cycles for all the patients enrolled in stages 1, 2 and 3
  Maximal Tolerated Dose/Recommended Phase 2 Dose (MTD/RP2D)
Stage 4: Progression Free Survival at 6 months | Day 1 of treatment until first documentation of disease progression or date of death, whichever comes first, assessed up to 6 months
  Progression Free Survival at 6 months will be estimated by the Kaplan-Meier method

SECONDARY OUTCOMES:
Overall Survival | 5 years
  Day 1 of treatment until death to calculate Median overall survival by the Kaplan-Meier method.
Progression Free Survival | 5 years
  Day 1 of treatment until first documentation of disease progression or death to calculate Median progression free survival by the Kaplan-Meier method.

CONTACTS AND LOCATIONS:
Locations (1):
- Duke University, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No